CLINICAL TRIAL: NCT05435456
Title: Effect of Strengthening and Relaxation Exercises on Musculoskeletal Pain, Anxiety, and Sleep Quality on Post-covid Symptoms
Brief Title: Effect of Exercise on Post-Covid Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Seda Saka, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ssaka7
Record Dates: First submitted 2022-06-26; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Performed strengthening and relaxation exercises 3 times a week for 8 weeks.
  Interventions: Other: Exercise
- Control Group (No Intervention): There is no intervention

INTERVENTIONS:
Other: Exercise — Strengthening and Relaxation Exercises
  Arms: Experimental Group

SUMMARY:
The study aimed to investigate the effects of strengthening and relaxation exercises on pain, anxiety, and sleep quality. 76 post-covid patients were randomized into experimental and control groups. Experimental group patients performed strengthening and relaxation exercises 3 times a week for 8 weeks. Control group patients did not perform any program. All participants were assessed with McGill Pain Scale short form (SFMPQ), short-form 36 (SF-36), Pittsburgh sleep quality index (PSQI) before and after the study.

DETAILED DESCRIPTION:
After COVID-19, musculoskeletal pain, anxiety, and sleep problems can continue. The study aimed to investigate the effects of strengthening and relaxation exercises on pain, anxiety, and sleep quality. The study was performed at Gaziosmanpaşa Education and Research Hospital with 76 post-covid patients that were randomized into experimental and control groups. Experimental group patients performed strengthening and relaxation exercises 3 times a week for 8 weeks. Control group patients did not perform any program. All participants were assessed with McGill Pain Scale short form (SFMPQ), short-form 36 (SF-36), and Pittsburgh sleep quality index (PSQI) before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* to be between the ages of 18-65
* to be diagnosed with Covid-19 in the last 3 months
* to have a negative PCR test, or to have completed the 14-day isolation period

Exclusion Criteria:

* have undergone surgery in the last 6 months
* have severe mental retardation that would prevent communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
McGill Pain Scale short form (SFMPQ) | at the enrollment and after the study
  It gives an information about the sensation, severity and effect of pain
Short-Form 36 (SF-36) | at the enrollment and after the study
  It asses general quality of life with 8 parameters
Pittsburg Sleep Quality Index | at the enrollment and after the study
  It asses sleep quality with 19 questions that each question scored between 0-3.
Beck Anxiety Scale | at the enrollment and after the study
  It asses anxiety levels with subjective and somatic factors

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PhD, Study Director — Haliç University
Locations (1):
- Gaziosmanpaşa Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Result] Liu K, Chen Y, Wu D, Lin R, Wang Z, Pan L. Effects of progressive muscle relaxation on anxiety and sleep quality in patients with COVID-19. Complement Ther Clin Pract. 2020 May;39:101132. doi: 10.1016/j.ctcp.2020.101132. Epub 2020 Mar 6. PMID 32379667